CLINICAL TRIAL: NCT06792565
Title: Hemofilters vs. Hemodialyzers: Impacts on Cytokine Removal During Cardiopulmonary Bypass in Pediatric Cardiac Surgery
Brief Title: Compare the Impact of Hemofilters and Hemodialyzers on Cytokine Removal During Cardiopulmonary Bypass in Pediatric Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alnas Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RHDIRB-NA-240823-01UC-NPO-N032
Record Dates: First submitted 2025-01-20; First posted 2025-01-24 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Cardio-pulmonary Bypass; Cytokine

STUDY DESIGN:
Intervention Model Description: compare impact of hemofilters and hemodialyzers on cytokine removal during cardiopulmonary bypass in pediatric cardiac surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hemodialyzers (Experimental): 20 patients
  Interventions: Device: hemodializer
- hemofilters (Active Comparator): 20 patients
  Interventions: Device: hemofilter

INTERVENTIONS:
Device: hemodializer — Fresenius Helixone FX5 (61346 Bad Homburg, Germany)
  Arms: hemodialyzers
Device: hemofilter — Medica (741036 Medolla, Italy)
  Arms: hemofilters

SUMMARY:
Cardiopulmonary bypass (CPB) allowed the correction of several congenital heart diseases such as intracardiac malformations, but it is well known that this is not a harmless procedure because it can lead to a systemic inflammatory response syndrome (SIRS), with activation of complement, cytokines, coagulation, and fibrinolysis pathways.

Due to economic causes, hemofilters became less available in low-resource countries, which forced perfusionists to use hemodialyzers instead during CPB. Preliminary data showed the potential safety of using hemodialyzers instead of hemofilters in Zero-balanced ultrafiltration.

The Objectives of the study This study aims to compare impact of hemofilters and hemodialyzers on cytokine removal during cardiopulmonary bypass in pediatric cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients who are undergoing elective cardiothoracic surgery which cardiopulmonary bypass will be conducted.
2. Age of patients from 1 year to 15 years.
3. CPB duration more than 60 minutes.

Exclusion Criteria:

1. Pediatric patients with known signs of sepsis.
2. Pediatric patients having had previous cardiothoracic surgery.
3. Preoperative renal failure.
4. Preoperative cardiogenic shock requiring the use of inotropes.
5. Preoperative lactate concentration > 2 mmol/L.

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-03-22 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
IL6 level as a proinflammatory cytokine | preoperatively after induction of anesthesia (T1), after removal of aorta cross clamp and before starting zero-balanced ultrafiltration (T2) and after coming off CPB (T3).

SECONDARY OUTCOMES:
Other proinflammatory cytokine | preoperatively after induction of anesthesia (T1), after removal of aorta cross clamp and before starting zero-balanced ultrafiltration (T2) and after coming off CPB (T3).
  IL1β, Lactate level

CONTACTS AND LOCATIONS:
Overall Officials: Amal F Rizk, MD, Study Director — Alnas Hospital
Locations (1):
- Alnas Hospital, Shubrā al Khaymah, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, Analytic Code